CLINICAL TRIAL: NCT06504810
Title: Effect of Light Level on Stress, Anxiety, Psychological Well-being in Pregnant Women: Randomized Placebo-controlled Study
Brief Title: Effect of Light Level on Stress, Anxiety, Psychological Well-being in Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1357
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Stress; Anxiety; Pregnant Women
MeSH Terms: conditions — Anxiety Disorders | interventions — Light

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator)
  Interventions: Other: light
- experimental group (Experimental)
  Interventions: Other: light

INTERVENTIONS:
Other: light — light level

SUMMARY:
To determine the effect of light level on stress, anxiety and psychological well-being in pregnant women. This research was planned as a single-blind, randomized controlled experimental type study by comparing separate groups as experiment-placebo control. Data will be collected using the Introductory Information Form, Psychological Well-Being Scale, Perceived Stress Scale (ASÖ/PSÖ-14), and State-Trait Anxiety Inventory (STAI). The effect of two different amounts of light on pregnant women will be evaluated.

DETAILED DESCRIPTION:
To determine the effect of light level on stress, anxiety and psychological well-being in pregnant women. This research was planned as a single-blind, randomized controlled experimental type study by comparing separate groups as experiment-placebo control. Data will be collected using the Introductory Information Form, Psychological Well-Being Scale, Perceived Stress Scale (ASÖ/PSÖ-14), and State-Trait Anxiety Inventory (STAI). The effect of two different amounts of light on pregnant women will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* being in the last trimester of pregnancy,
* volunteering.

Exclusion Criteria:

* Having any problems that prevent you from communicating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-07-26 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
stress | 1 day
  stress scale

SECONDARY OUTCOMES:
anxiety | 1 day
  anxiety scale